CLINICAL TRIAL: NCT07365371
Title: A Prospective, Multicenter, Open-label, Randomized Clinical Trial to Evaluate the Efficacy, Durability, and Safety of Aflibercept 8mg in Different Treatment Regimens in Chinese Patients With Polypoidal Choroidal Vasculopathy (PCV)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Xiaodong Sun, Vice president of Shanghai General Hospital, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23106
Record Dates: First submitted 2025-12-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Polypoidal Choroidal Vasculopathy (PCV); Neovascular Age Related Macular Degeneration (AMD)
Keywords: Polypoidal Choroidal Vasculopathy (PCV); Neovascular age related macular degeneration (AMD); Aflibercept 8mg
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Other): All enrolled patients meeting eligibility will receive intravitreal aflibercept 8 mg loading doses (3 initial monthly doses). Subsequent reinjections will be given according to the changes in patients' disease activity. If no retreatment criteria are met, no additional injections will be given, and patients will undergo follow-up examinations (including ETDRS visual acuity, findus photography, OCT-A and SD-OCT) every 4 weeks until week 48. Patients will return to the Clinical Research Unit (CRU) for an end-of-study (EOS) visit at week 52.
  Interventions: Drug: Aflibercept Intravitreous Injection
- Arm B (Other): All enrolled patients meeting eligibility will receive intravitreal aflibercept 8 mg loading doses (3 initial monthly doses). All patients in this group will undergo an examination at week 12, including ETDRS visual acuity, fundus photography, OCT-A and SD-OCT. Subsequent treatment regime will depend on disease activity. If disease is considered inactive, the next dose will occur at week 16 (8 week interval from last dose at week 8) and subsequent dose and visit will be extended by 4 weeks up to a maximum interval of 20 weeks and minimum interval of 8 weeks between treatments if disease remains quiescent. If signs of activity are noted at any visit point, visit interval will be reduced by 4 weeks. The last dose will be administered no later than week 48. Patients will return to the CRU for an EOS visit at week 52.
  Interventions: Drug: Aflibercept Intravitreous Injection

INTERVENTIONS:
Drug: Aflibercept Intravitreous Injection — Patients will be given IVT injection(s) of IMP using standard injection techniques.

SUMMARY:
The goal of this clinical trial is to investigate the efficacy, durability, and safety of aflibercept 8 mg in treating Polypoidal Choroidal Vasculopathy (PCV) in Chinese naive patients. The main questions it aims to answer are:

1. What is the change in Best Corrected Visual Acuity (BCVA) at Week 52 from baseline in different treatment regimens?
2. What proportion of patients achieve sustained disease control after receiving the loading dose?

Participants will:

* Receive intravitreal aflibercept 8 mg loading doses (3 initial monthly doses).
* In Arm A:
* Undergo reinjections based on disease activity, with follow-up examinations every 4 weeks until week 48.
* Return for an end-of-study visit at week 52.
* In Arm B:
* Undergo an examination at week 12 and subsequent treatments based on disease activity, with a maximum interval of 20 weeks and a minimum interval of 8 weeks between doses if the disease remains inactive.
* Return for an end-of-study visit at week 52.

This study will assess the efficacy, safety and durability of aflibercept 8mg in these 2 regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fully understand the content, process, and possible AE of the study and capable of giving written informed consent form.
* Male or female, age ≥ 50 years, at the time of signing the informed consent form.
* Women of childbearing potential (WOCBP) must agree to practice a double method of contraception of a medically acceptable method of contraception with an annual failure rate of less than 1% (see Appendix 1) with a barrier contraceptive (such as condom) during the study and for 4 months after discontinuation of study treatment. Women are considered not of childbearing potential if they are surgically sterile (i.e., hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) or > 1 year postmenopausal. WOCBP must have negative results of pregnancy test at screening and must not be pregnant, breast feeding, lactating, or planning to become pregnant, breast feed or donate ova during the study and for 4 months after discontinuation of study treatment.
* All male participants with female partners of childbearing potential must agree to practice a double method of contraception of a medically acceptable method of contraception with an annual failure rate of less than 1% (see Appendix 1) with a barrier contraceptive (such as condom), and must agree to abstain from sperm donation during and for 4 months after participation in the study.
* Ocular Inclusion Criteria for Study Eye: Sufficiently clear ocular media and adequate pupillary dilatation to allow acquisition of good quality retinal images to confirm diagnosis.
* Ocular Inclusion Criteria for Study Eye: Confirmed diagnosis, by the investigator, of symptomatic macular PCV defined by the following: a. Active macular polypoidal lesions shown by ICGA, AND presence of CNV involving the macula area within the 6.0 mm ETDRS zone as identified by the investigator using multimodal images. b. BCVA scores of 78~24 ETDRS letters, inclusive (20/32 to 20/320 approximate Snellen equivalent), using the ETDRS protocol and assessed at the initial testing distance of 4 meters on study Day 1 Note: If both eyes meet the inclusion criteria, the eye with the worst visual acuity (VA) at the screening visit will be designated as the study eye. If both eyes have the same VA, the Investigator and patient will determine the study eye.

Exclusion Criteria:

* Treatment with investigational therapy (anti-VEGF, corticosteroid, laser photocoagulation, panretinal or macular, and PDT) or approved medications for PCV treatment prior to initiation of study treatment on study Day 1.
* Allergy or hypersensitivity to any of the compounds/excipients in the study interventions formulations.
* Uncontrolled blood pressure (defined as systolic >160 mmHg or diastolic >95 mmHg). Participants may be treated with up to 3 agents known to have anti-hypertensive effects for arterial hypertension to achieve adequate blood pressure control. This limit applies to drugs that could be used to treat hypertension even if their primary indication in the participant was not for blood pressure control. Any recent changes in medications known to affect blood pressure need to be stable for 12 weeks prior to screening.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, might affect interpretation of the results of the study, or renders the participant at high risk for treatment complications.
* Any other conditions that the Investigator considers may affect the patients' informed consent or adherence to the study protocol, completion of the test according to the study procedure, or the patients' participation in the test may affect the test results or their own safety.
* Pregnant or breastfeeding.
* Ocular Exclusion Criteria for Study Eye: Any history or presence of macular pathology unrelated to PCV affecting vision or contributing to the presence of macular hemorrhage, IRF, or SRF.
* Ocular Exclusion Criteria for Study Eye: Retinal pigment epithelial tear involving the macula on study Day 1.
* Ocular Exclusion Criteria for Study Eye: On FA/ fundus photograph (FP): a. Subretinal hemorrhage of >4 macular photocoagulation study disc area and/or that involves the fovea b. Fibrosis or atrophy of >50% of the total lesion area and/or that involves the fovea
* Ocular Exclusion Criteria for Study Eye: Any concurrent intraocular condition (e.g., amblyopia, aphakia, retinal detachment, cataract, DR or maculopathy, or epiretinal membrane with traction) that, in the opinion of the investigator, could either reduce the potential for visual improvement or require medical or surgical intervention during the study a. Current vitreous hemorrhage on study Day 1 b. Uncontrolled glaucoma c. Any cataract surgery or treatment for complications of cataract surgery with steroids or YAG laser capsulotomy within 3 months prior to study Day 1 d. Any other intraocular surgery (e.g., pars plana vitrectomy, glaucoma surgery, corneal transplant, or radiotherapy) e. Prior periocular pharmacological or IVT treatment (including anti-VEGF medication) for other retinal diseases • Evidence of infectious blepharitis, keratitis, scleritis, or conjunctivitis in either eye within 4 weeks of the screening visit f. Any intraocular inflammation/infection in either eye within 12 weeks of the screening visit g. History of idiopathic or autoimmune uveitis in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) change at Week 52 after baseline in different treatment regimens. | up to 52 Weeks
  BCVA (study eye and the fellow eye) examination

SECONDARY OUTCOMES:
Percentage of patients gaining >15, >10, or ≥5 letters in BCVA after baseline | up to 52 Weeks
  BCVA (study eye and the fellow eye) examination
Percentage of patients achieving complete polypoidal lesion regression at Weeks 52 | up to 52 Weeks
  SD-OCT Spectral Domain Optical Coherence Tomography, FA Fluorescein Angiography, ICGA Indocyanine Green Angiography, OCT-A Optical Coherence Tomography Angiography, FP Fundus Photography examinations
Percentage of patients with no active polypoidal lesion at Week 52 | up to 52 Weeks
  SD-OCT Spectral Domain Optical Coherence Tomography, FA Fluorescein Angiography, ICGA Indocyanine Green Angiography, OCT-A Optical Coherence Tomography Angiography, FP Fundus Photography examinations
Change from baseline in central subfield thickness (CST) at Week 12 and 52. | up to 12 and 52 Weeks
  SD-OCT Spectral Domain Optical Coherence Tomography examination
BCVA change from baseline at Week 12 | up to 12 Weeks
  BCVA (study eye and the fellow eye) examination
Percentage of patients achieving Q8W, Q12W, and Q16W treatment intervals at Week 52 in Arm B. | up to 52 Weeks
  Calculating the ratio
Percentage of patients achieving Q20W of last assigned interval at Week 52 in Arm B. | up to 52 Weeks
  Calculating the ratio
Percentage of patients achieving ≥12-week, ≥16-week and ≥20-week treatment intervals after completing loading doses in Arm A. | up to 52 Weeks
  Calculating the ratio
Total number of intravitreal injections administered through Week 52 in both arms. | up to 52 Weeks
  Counting
Incidence and severity of ocular & non-ocular adverse events. | up to 52 Weeks
  Recording of adverse events

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, CMU, Beijing, Beijing Municipality
  - The Second People's Hospital Of Foshan, Foshan, Guangdong
  - The First Affiliated Hospital Of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Renmin Hospital Of Wuhan University, Wuhan, Hubei
  - Jiangsu Province Hospital , The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Eye Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Norman Bethune Hospital Of Jilin University, Jilin, Jilin
  - Xi' AN No.1 Hospital, Xi'an, Shaanxi
  - The First People's Hospital Of Xianyang, Xianyang, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Affiliated Hospital Of Shandong Second Medical University, Weifang, Shandong
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Eye Hospital, Taiyuan, Shanxi
  - Tianjin Eye Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jiaxing Hospital of T.C.M, Jiaxing, Zhejiang
  - Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No